CLINICAL TRIAL: NCT06280196
Title: A Phase I/III, Multi-center, Randomized, Double-blind Study of BAT3306 Plus Chemotherapy Versus Keytruda® Plus Chemotherapy to Evaluate Pharmacokinetics, Efficacy, and Safety in Participants With Stage IV Non-squamous Non-small Cell Lung Cancer.
Brief Title: A Study to Evaluate PK, Efficacy, and Safety of BAT3306 Plus Chemo and Compare With Keytruda®(EU/US) in Participants With IV nqNSCLC
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The new regulatory developments have led us to conclude that a Phase 3 study is no longer necessary for the development and approval of BAT3306. As such, to ensure effective use of clinical resources, we are terminating this study.
Sponsor: Bio-Thera Solutions (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BAT-3306-002-CR
Record Dates: First submitted 2024-02-04; First posted 2024-02-28 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-12

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — pembrolizumab; Pemetrexed; Carboplatin

STUDY DESIGN:
Intervention Model Description: double-blind, randomized
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- BAT3306 (Experimental): 25 mg/mL concentrate for solution for infusion.200 mg on Day 1 of each 21-day cycle
  Interventions: Drug: BAT3306; Drug: Pemetrexed; Drug: Carboplatin
- EU-Keytruda® arm (Active Comparator): 25 mg/mL concentrate for solution for infusion.200 mg on Day 1 of each 21-day cycle
  Interventions: Drug: EU-Keytruda®; Drug: Pemetrexed; Drug: Carboplatin
- US-Keytruda® arm (Active Comparator): 25 mg/mL concentrate for solution for infusion. 200 mg on Day 1 of each 21-day cycle
  Interventions: Drug: US-Keytruda®; Drug: Pemetrexed; Drug: Carboplatin

INTERVENTIONS:
Drug: BAT3306 — One vial of 4 mL of concentrate contains 100 mg of BAT3306
  Other Names: Pembrolizumab Injection
  Arms: BAT3306
Drug: EU-Keytruda® — One vial of 4 mL of concentrate contains 100 mg of pembrolizumab
  Other Names: Pembrolizumab Injection
  Arms: EU-Keytruda® arm
Drug: US-Keytruda® — One vial of 4 mL of concentrate contains 100 mg of pembrolizumab
  Other Names: Pembrolizumab Injection
  Arms: US-Keytruda® arm
Drug: Pemetrexed — 500 mg/m2 on Day 1 of each 21-day cycle of the study
  Other Names: Pemetrexed Fresenius Kabi
Drug: Carboplatin — Target AUC of 5 mg/mL/min on Day 1 of each 21-day cycle up to 4 cycles
  Other Names: Carboplatin Kabi

SUMMARY:
To compare the pairwise PK similarities between BAT3306, EU-Keytruda, and US-Keytruda, all administered with pemetrexed and carboplatin.

DETAILED DESCRIPTION:
This is a multi-center, double-blind, randomized study that includes PK and clinical equivalence comparisons, aimed at comparing BAT3306 with Keytruda® in previously untreated participants with Stage IV nsNSCLC.

ELIGIBILITY:
Inclusion Criteria:

* Participants are eligible to be included in the study only if all the following criteria are met:

  1. Male or female, age ≥18 years on the day of signing informed consent.
  2. Participants are able to give voluntary informed consent and understand the study and are willing to follow and complete all the test procedures.
  3. Life expectancy ≥3 months, per the investigator's evaluation.
  4. Eastern Cooperative Oncology Group (ECOG) performance status ≤1.
  5. Histologically/cytologically confirmed diagnosis of Stage IV (AJCC 8th edition) nsNSCLC.
  6. Tumors without EGFR mutation/ROS1 rearrangement /ALK rearrangement.

Exclusion Criteria:

* Participant must be excluded from participating in the study if the participant:

  1. Is pregnant or a nursing female.
  2. Has predominantly squamous cell histology NSCLC. Mixed tumors will be categorized by the predominant cell type; if small cell elements are present, the participant is ineligible.
  3. Is currently participating and receiving an investigational agent or has participated in a study of an investigational agent and received an investigational agent or used an investigational device within 4 weeks prior to administration of the first dose of study intervention.
  4. Before the first dose of study intervention:

     * Had received prior systemic antineoplastic chemotherapy and targeted, biological therapy
     * Had prior treatment with any other anti-PD-1, PD-L1 or PD-L2 agent or an antibody targeting other immuno-regulatory receptors or mechanisms. Examples of such antibodies include (but are not limited to) antibodies against TIGIT, IDO, PD-L1, CTLA-4, and LAG3.
     * Has participated in any other BAT3306 study and has been treated with BAT3306.
     * Had major surgery <3 weeks prior to first dose
     * Received radiation therapy to the lung that is > 30 Gy within 6 months of the first dose of study intervention.
     * Completed palliative radiotherapy within 14 days of the first dose of study intervention.
  5. Is expected to require any other form of antineoplastic therapy while participating in the study. and so on

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2024-07-19 (Actual); Primary Completion 2025-07-30 (Actual); Study Completion 2025-07-30 (Actual)

PRIMARY OUTCOMES:
clinical equivalence | Week 3,5,7,9,12,15,EOT
  To compare the efficacy of BAT3306 and pooled EU-Keytruda® and US-Keytruda® given with chemotherapy as first line treatment using ORR assessed by BIRC to show clinical equivalence in participants with nsNSCLC. Confirmed best overall tumor response rate as assessed by BIRC according to RECIST Version 1.1 (tumor assessments after initiation of a new anti-cancer treatment are excluded)

SECONDARY OUTCOMES:
safety of BAT3306 | From signed ICF to 90days after the last drug administration
  The Investigator and any qualified designees are responsible for detecting, documenting, and reporting events that meet the definition of an AE or SAE and remain responsible for following up AE that are serious, considered related to the study intervention or the study, or that caused the participant to discontinue the study.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaorong Dong, Dr., Principal Investigator — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Locations (1):
- Union Hospital Tongji Medical College Huazhong University of Science & Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No